CLINICAL TRIAL: NCT03171883
Title: The Value of Ultrasound in the Diagnosis of Supraspinatus Muscle Tears
Brief Title: Ultrasound of Supraspinatus Muscle Tears
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherry Ayad, principal investigator, Assiut University
Other Study IDs: USSPMT
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Supraspinatus Tear or Rupture, Not Specified as Traumatic
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The supraspinatus is a relatively small muscle of the upper back that runs from the supraspinatus fossa superior portion of the scapula to the greater tubercle of the humerus. It is one of the four rotator cuff muscles and also abducts the arm at the shoulder. A supraspinatus tear is a tear or rupture of the tendon of the supraspinatus muscle.

DETAILED DESCRIPTION:
Many pathological conditions as trauma (whether acute or chronic), inflammation or instability may cause supraspinatus muscle disease which is one of the commonest cause of shoulder pain and malfunction.

Supraspinatus muscle failure usually results from tendinopathy that transforms from partial to full thickness tears.

Basically shoulder impingement is a clinical diagnosis. The role of imaging in such condition is to identify the causal factors as well as to detect the involvement of tendon injuries and its extension as tears of the cuff muscles is difficult to be identified clinically.

The decision making in the treatment of the supraspinatus muscle tears relies mainly upon the correct diagnosis of the type and extent of the tear. According to the diagnosis whether conservative or surgical treatment is chosen, even the type of the surgical intervention (open or arthroscopic) would differ according to the diagnosis.

In addition identifying the extent of tendons retraction and the condition of the ruptured edges, as well as the quality of the muscle itself influences the management policy.

To evaluate the painful shoulder a variety of imaging tests have been used; yet, for diagnosing a supraspinatus muscle tear the standard imaging modalities such as unenhanced magnetic resonance imaging, indirect and direct magnetic resonant arthrography, and ultrasound are used.

US of the shoulder is utilized increasingly in healthcare settings to assess the integrity of the supraspinatus muscle. It is a non-invasive examination with practically no side effects. It is beneficial in the dynamic examination of the tendon during movement of the shoulder .

ELIGIBILITY:
Inclusion Criteria:

* patients of different age groups presented with clinical diagnosis department of shoulder impingement and diagnosed by magnetic resonance imaging as supraspinatus

Exclusion Criteria:

* patients with previous shoulder surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of different age groups presented with clinical diagnosis of shoulder impingement
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Patients diagnosed as supraspinatus lesions by ultrasound | 2 years
  Evaluation the effectiveness of ultrasound in the assessment of supraspinatus muscle tears compared with results of shoulder arthroscopy as a gold standard method.

REFERENCES:
- [Background] Lewis JS. Rotator cuff tendinopathy: a model for the continuum of pathology and related management. Br J Sports Med. 2010 Oct;44(13):918-23. doi: 10.1136/bjsm.2008.054817. Epub 2009 Apr 12. PMID 19364757
- [Background] Fotiadou AN, Vlychou M, Papadopoulos P, Karataglis DS, Palladas P, Fezoulidis IV. Ultrasonography of symptomatic rotator cuff tears compared with MR imaging and surgery. Eur J Radiol. 2008 Oct;68(1):174-9. doi: 10.1016/j.ejrad.2007.11.002. Epub 2007 Dec 21. PMID 18160242
- [Background] Whiting P, Rutjes AW, Reitsma JB, Bossuyt PM, Kleijnen J. The development of QUADAS: a tool for the quality assessment of studies of diagnostic accuracy included in systematic reviews. BMC Med Res Methodol. 2003 Nov 10;3:25. doi: 10.1186/1471-2288-3-25. PMID 14606960
- [Background] Le Corroller T, Cohen M, Aswad R, Pauly V, Champsaur P. Sonography of the painful shoulder: role of the operator's experience. Skeletal Radiol. 2008 Nov;37(11):979-86. doi: 10.1007/s00256-008-0539-z. Epub 2008 Jul 24. PMID 18651142